CLINICAL TRIAL: NCT06435845
Title: A Phase 2, Multicenter, Open-label Study to Evaluate the Pharmacokinetics and Safety of RLYB212 in Pregnant Women at Higher Risk for HPA-1a Alloimmunization
Brief Title: Phase 2 Study on the Pharmacokinetics and Safety of RLYB212 in Pregnant Women at Higher Risk for HPA-1a Alloimmunization
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated early by the sponsor due to insufficient drug exposure to achieve the intended therapeutic effect.
Sponsor: Rallybio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IPA2202; 2024-512651-20-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-21; First posted 2024-05-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Fetal and Neonatal Alloimmune Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia, Neonatal Alloimmune

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- RLYB212 (Experimental): RLYB212 Subcutaneous injection
  Interventions: Drug: Anti-(integrin beta-3) human monoclonal antibody

INTERVENTIONS:
Drug: Anti-(integrin beta-3) human monoclonal antibody — human monoclonal anti-human platelet antigen (HPA)-1a immunoglobulin G antibody
  Other Names: RLYB212

SUMMARY:
The purpose of this Phase 2 study is to assess the pharmacokinetics (PK) and safety of RLYB212 in HPA-1b/b pregnant women at higher risk for HPA-1a alloimmunization and FNAIT.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, multicenter study of RLYB212 in HPA-1b/b pregnant participants at higher risk for the occurrence of HPA-1a alloimmunization and FNAIT. A laboratory testing paradigm will be applied at screening to identify women at higher risk for HPA-1a alloimmunization. Study IPA2202 is comprised of three phases: a two-part screening phase, an antenatal treatment phase, and a postpartum follow-up phase. Study duration for each participant is anticipated to be ~44 weeks, inclusive of the screening visits through the Week 10 postpartum visit.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women who present at Gestational Week 6 or after and confirmed to be: HPA-1b/b (HPA-1a negative), HLA-DRB3*01:01 positive, Anti-HPA-1a alloantibody negative, Carrying an HPA-1a/b (HPA-1a positive) fetus

Exclusion Criteria:

* Prior history of HPA-1a related fetal and neonatal alloimmune thrombocytopenia
* Multiple pregnancy (more than 1 fetus)
* Prior history of platelet transfusion or other blood transfusions
* Known sensitivity and/or immediate hypersensitivity to any components of RLYB212 or its formulation
* Any co-morbid medical or obstetric condition(s), laboratory abnormality, concomitant treatment, or other reason that, in the investigator's opinion, could adversely affect the safety of the participant and/or fetus, impair the assessment of study results, or preclude compliance with the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 1 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with treatment related adverse events as defined by CTCAE 5.0 | Approx. Gestational Week (GW) <16, 16, 18, 20, 24, 26, 28, 30, 32, 34, 36, 38; at birth (~40), Post Partum (PP) Week 4, 10 week
Maternal exposure to RLYB212 as measured in serum | Approx. GW 16, 18, 20, 24, 26, 28, 30, 32, 34, 36, 38, at birth (~40), PP Week 4

SECONDARY OUTCOMES:
Neonatal exposure to RLYB212 as measured in cord blood | At birth (~GW 40)
Number of HPA-1a positive neonates with treatment related adverse events as defined by CTCAE v5.0 | At birth (~GW 40), Approx. PP Week 4
Anti-RLYB212 antibodies as measured in serum | Approx. GW 16, 20, 24, 28, 32, 36, at birth (~40), PP Week 4
Pregnancy Outcomes: incidence of live births, spontaneous abortions, elective abortions, still births or premature births | At birth (~GW 40)
Frequency of Neonatal Thrombocytopenia as measured by platelet count within 72 hours of delivery | At birth (~GW 40)
Frequency of HPA-1a Alloimmunization as measured by anti-HPA-1a alloantibodies | Approx. PP Week 10
Neonatal Outcomes: general health and overall status as defined by absolute values and percentiles | 4-6 weeks following delivery

CONTACTS AND LOCATIONS:
Locations (3):
- Leids Universitair Medisch Centrum, Leiden, South Holland, Netherlands
- Oslo University Hospital- Ullevål, Oslo, Oslo County, Norway
- Södersjukhuset, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT06435845/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT06435845/SAP_001.pdf